CLINICAL TRIAL: NCT02939755
Title: Collaborative Care Intervention for Cancer Patients and Their Family Caregivers
Brief Title: Web-based Collaborative Care Intervention Study
Acronym: WBCCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Director and Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY19050065
Record Dates: First submitted 2016-10-14; First posted 2016-10-20 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Depression; Fatigue; Pain
Keywords: Collaborative care intervention; Cancer; Depression; Palliative care; Quality of life; Fatigue; Pain
MeSH Terms: conditions — Neoplasms; Depression; Fatigue; Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped collaborative care intervention (Experimental): The 'Stepped Collaborative Care Intervention' includes at least biweekly contact from a care coordinator by phone and face to face visits occurring approximately every 2 months, and 24 hour 7 day a week access to a website that was specifically designed during the pilot study for advanced cancer patients from socioeconomically disadvantaged backgrounds.
  Interventions: Behavioral: Stepped collaborative care intervention
- Enhanced Usual Care (Active Comparator): Patients randomized to the 'Enhanced Usual Care' arm receive their usual care from their medical team. However, if the patient scores in the clinical range on one or more of the three symptoms s/he will receive education about the symptom and be referred to the appropriate health care provider for further treatment in their community. The care coordinator will follow up with the patient after 3 weeks to assess barriers to treatment and assist further with accessing treatment if needed.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Stepped collaborative care intervention — Using website that was specifically designed for advanced cancer patient, collaborative with treatment from health professional
  Other Names: treatment
  Arms: Stepped collaborative care intervention
Behavioral: Enhanced Usual Care — usual care from health providers
  Other Names: control
  Arms: Enhanced Usual Care

SUMMARY:
To test the efficacy of a web-based stepped collaborative care intervention to reduce symptoms of depression, pain, and fatigue and improve health-related quality of life (HRQL) in advanced cancer patients and to reduce stress and depression, and fewer CVD risk factors in caregivers.

DETAILED DESCRIPTION:
The investigators will enroll patients at two UPMC sites: Montefiore Hospital, an academic medical center, and Passavant Hospital, a community based hospital. Based on our sample size estimate the investigators will have at least 364 patients and caregivers with complete data at 12 months follow up.

The patient and caregiver will be randomly assigned to one of two arms (intervention versus enhanced usual care) stratified by gender and vessel invasion. Because these factors are the two most robust prognostic factors in this patient population. At 6 and 12 months after enrollment, follow-up questionnaires and blood draws will be performed for patients and caregivers.

The stepped WBCC intervention includes at least biweekly contact from a care coordinator by phone and face to face visits occurring approximately every 2 months, and 24 hour 7 day a week access to a website. Patients randomized to the "enhanced usual care" arm receive their usual care from their medical team. However, if the patient scores in the clinical range on one or more of the three symptoms s/he will receive education about the symptom and be referred to the appropriate health care provider for further treatment in their community. The care coordinator will follow up with the patient after 3 weeks to assess barriers to treatment and assist further with accessing treatment if needed.

Intervention fidelity (e.g., consistency across care coordinators) will be reduced by requiring the care coordinators to follow a 300 page manual and providing standardized training by the PI who is a clinical psychologist. Dr. Steel (PI) has received training and certification from the American Psycho-Oncology Society in the design and analysis of psycho-oncology clinical trials and intervention fidelity. The study investigators will not prescribe any medications but rather make recommendations to the patient's oncologist, PCP, psychiatrist, or pain management specialist who will be free to accept or reject the recommendations by the study team. Medication type, dosage, and adherence to medication (e.g., self-report and pharmacy refills) will be recorded for patients in the WBCC intervention and enhanced usual care arms.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* biopsy and/or radiograph proven diagnosis of hepatocellular carcinoma,cholangiocarcinoma, gallbladder carcinoma or breast, ovarian, or colorectal cancer with liver metastases with a life expectancy of at least one year;
* age >21 years;
* no evidence of thought disorder, delusions, or active suicidal ideation is observed or reported.

Caregivers:

* a spouse or cohabitating intimate partner of an advanced cancer patient being evaluated at the UPMC's Liver Cancer Center and
* age >21 years

Exclusion Criteria:

Patients:

* age < 21 years,
* lack of fluency in English,
* evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

Caregivers:

* lack of fluency in English; and
* evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | change from baseline at 6 and 12 months
  Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire

SECONDARY OUTCOMES:
serum Interleukin (IL)-6,(mg/L) | change from baseline at 6 months and 12 months
  Blood sample collection and process
serum Cancer Antigen 19-9 (u/ml) | change from baseline at 6 months and 12 months
  Blood sample collection and process
serum carcinoembryonic antigen (u/ml) | change from baseline at 6 months and 12 months
  Blood sample collection and process
serum Alpha feta protein (u/ml) | change from baseline at 6 months and 12 months
  Blood sample collection and process
Caregivers' stress | change from baseline at 6 and 12 months
  Caregiver Quality of Life Scale- Cancer, Perceived Stress Scale
Caregivers' depression | change from baseline at 6 and 12 months
  Center for Epidemiological Studies- Depression
dyadic adjustment | change from baseline at 6 and 12 months
  Dyadic Adjustment Scale
Caregiver's blood pressure | change from baseline at 6 and 12 months
  Blood pressure readings
Caregiver's Body Mass Index | change from baseline at 6 and 12 months
  Caregiver's height and weight calculations in inches and pounds using BMI calculator
Caregiver's serum Interleukin-6 | change from baseline at 6 and 12 months
  Blood sample collection and process
Caregiver's metabolic syndrome | change from baseline at 6 and 12 months
  The caregiver meets or does not meet the American Heart Association criteria for metabolic syndrome
Depression | change from baseline at 6 and 12 months
  Center for Epidemiological Studies- Depression
Fatigue | change from baseline at 6 and 12 months
  Functional Assessment of Cancer Therapy -fatigue
Pain level | change from baseline at 6 and 12 months
  Brief Pain Inventory
serum Interleukin IL-1beta,(mg/L) | change from baseline at 6 and 12 months
  cytokine
serum Tumor necrosis factor-alpha ((mg/L) | change from baseline at 6 and 12 months
  cytokine
serum Inteferon-gamma ((mg/L) | change from baseline at 6 and 12 months
  cytokine

OTHER OUTCOMES:
Health care utilization | 1 year
  Emergency Room visits, 30- and 90-day readmissions, length of stay in the hospital.
Health care costs | 12 months
  activity based costs

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Steel, PhD, Principal Investigator — UPMC Departemnt of Surgery
Locations (7):
- United States (7):
  - UPMC East, Monroeville, Pennsylvania
  - The University of Pittsburgh's Medical Center Passavant Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Mercy, Pittsburgh, Pennsylvania
  - University of Pittsburgh's Medical Center Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Horizen, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-Identified Data may be shared with investigators who request data from the Primary Investigator
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the end of the study for up to one year.
Access Criteria: Appropriate investigator credentials (MD, PhD) and request, and for up to one year after study completion

REFERENCES:
- [Derived] Diamantis GN, Kim Y, Ofori-Atta Z, Devine L, Antoni MH, Reyes V, Johnson J, Kiefer G, Jiang Y, Zandberg DP, Nilsen M, Tohme S, Geller DA, Steel JL. The interdependence of depressive symptoms and sleep in dyads affected by cancer. Health Psychol. 2025 Apr;44(4):391-400. doi: 10.1037/hea0001449. Epub 2024 Nov 25. PMID 39585770
- [Derived] Steel JL, George CJ, Terhorst L, Yabes JG, Reyes V, Zandberg DP, Nilsen M, Kiefer G, Johnson J, Marsh C, Bierenbaum J, Tageja N, Krauze M, VanderWeele R, Goel G, Ramineni G, Antoni M, Vodovotz Y, Walker J, Tohme S, Billiar T, Geller DA. Patient, family caregiver, and economic outcomes of an integrated screening and novel stepped collaborative care intervention in the oncology setting in the USA (CARES): a randomised, parallel, phase 3 trial. Lancet. 2024 Apr 6;403(10434):1351-1361. doi: 10.1016/S0140-6736(24)00015-1. Epub 2024 Mar 12. PMID 38490230
- [Derived] Steel JL, Amin A, Peyser T, Olejniczak D, Antoni M, Carney M, Tillman E, Hecht CL, Pandya N, Miceli J, Reyes V, Nilsen M, Johnson J, Kiefer G, Pappu B, Zandberg DP, Geller DA. The benefits and consequences of the COVID-19 pandemic for patients diagnosed with cancer and their family caregivers. Psychooncology. 2022 Jun;31(6):1003-1012. doi: 10.1002/pon.5891. Epub 2022 Feb 1. PMID 35083809
- [Derived] Steel JL, Reyes V, Zandberg DP, Nilsen M, Terhorst L, Richards G, Pappu B, Kiefer G, Johnson J, Antoni M, Vodovotz Y, Spring M, Walker J, Geller DA. The next generation of collaborative care: The design of a novel web-based stepped collaborative care intervention delivered via telemedicine for people diagnosed with cancer. Contemp Clin Trials. 2021 Jun;105:106295. doi: 10.1016/j.cct.2021.106295. Epub 2021 Feb 5. PMID 33556589